CLINICAL TRIAL: NCT05057858
Title: Pharmacology of TDF-FTC Pre-exposure Prophylaxis in Kenyan Cisgender Women
Brief Title: The Women TDF-FTC Benchmark Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Colorado, Denver (Other); Kenya Medical Research Institute (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Assistant Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00011136; R01AI155086 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: Pre-exposure Prophylaxis; HIV; Kenya
MeSH Terms: conditions — HIV Infections | interventions — Racivir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Perfect Adherence (Experimental): Cisgender women will receive a single tablet of co-formulated 300 mg TDF/ 200mg FTC once daily (7 doses per week).
  Interventions: Drug: co-formulated 300 mg TDF/ 200mg FTC
- Moderate Adherence (Experimental): Cisgender women will receive a single tablet of co-formulated 300 mg TDF/ 200mg FTC tablet 4 times per week (Monday, Tuesday, Thursday, Friday)
  Interventions: Drug: co-formulated 300 mg TDF/ 200mg FTC
- Poor Adherence (Experimental): Cisgender women will receive a single tablet of co-formulated 300 mg TDF/ 200mg FTC tablet twice per week(Monday and Tuesday)
  Interventions: Drug: co-formulated 300 mg TDF/ 200mg FTC

INTERVENTIONS:
Drug: co-formulated 300 mg TDF/ 200mg FTC — Participants will be randomized into 1 of 3 groups to receive a controlled number of doses of a single tablet co-formulated 300 mg TDF/ 200mg FTC
  Other Names: Truvada

SUMMARY:
The study seeks to define the expected blood levels of pre-exposure prophylaxis (PrEP) medications (tenofovir) for cisgender women taking directly observed oral PrEP therapy to understand the frequency of PrEP dosing associated with HIV protection in cisgender women. Cisgender women will be randomly assigned to receive varying frequency of weekly PrEP doses and followed for up to 16 weeks. The study will also investigate how pregnancy affects the expected blood levels to help define optimal dosing of PrEP for HIV prevention during pregnancy.

DETAILED DESCRIPTION:
This is an open-label, randomized, three-arm, directly observed therapy study. HIV-uninfected non-pregnant cisgender women at low risk for HIV will be randomly assigned to 1 of 3 dosing frequencies of directly observed therapy (DOT) Tenofovir Disoproxil Fumarate/Emtricitabine (TDF/FTC) PrEP to help differentiate poor and modest from perfect dosing. An additional contemporaneous cohort of pregnant to receive daily dosing will also be recruited to evaluate the impact of pregnancy on blood and cellular drug levels. Drug concentrations in blood, vaginal fluid, and tissue will be measured during the study. The primary objectives of the study are:

1. To define the cisgender women-specific expected blood concentrations and dose-proportionality for Tenofovir-diphosphate (TFV-DP) in dried blood spots (DBS) and Peripheral Blood Mononuclear Cells(PBMCs) using directly observed TDF/FTC therapy at 2, 4, 7 doses per week.
2. To establish a model to predict adherence rate to TDF/FTC by level of TFV-DP in DBS for cisgender women. HIV-uninfected non-pregnant cisgender women will be randomly assigned to 1 of 3 dosing frequencies of directly observed therapy (DOT) TDF/FTC PrEP: 2, 4, or 7 doses/week to help differentiate poor and modest from perfect adherence.

The study will be the first to define TDF-PrEP adherence-blood concentration thresholds for African cisgender women, a priority population for HIV prevention. The findings will guide accurate interpretation of adherence and success of PrEP programs in cisgender women. This data will also help guide decisions on optimal PrEP dosing for HIV at-risk pregnant cisgender women in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤30 years old
* Willing to undergo urine pregnancy tests
* Has understood the information provided and has provided written informed consent before any study-related procedures are performed.
* HIV uninfected based on negative HIV rapid tests, according to Kenyan national algorithm
* Normal renal function (estimated glomerular filtration rate >60 mL/min)
* Hepatitis B surface Ag negative
* No active clinically significant medical or psychiatric conditions that would interfere with study participation
* Lack of severe anemia
* Willing to use DOT and come to clinic frequently for DOT PrEP for at least 8 weeks
* Willing to have home visits for follow up
* Has access to an active smartphone to allow off-site observation of dosing if unable to come to the clinic or as determined by the study staff, the participant resides in close location to clinic to permit home visit if unable to come to the clinic. i.e., potential participants without a smartphone may be enrolled in the study if investigator determines that the participant resides within reasonable distance from the clinic that would permit home visit id the participant misses their visit.
* Intention to stay within the study site's catchment area for at least 8 weeks.
* Resides or works in catchment area with high speed internet coverage to permit video streaming

Specific for non-pregnant cisgender women cohort

* Not pregnant or breast feeding
* At low risk for HIV. In Kenya, national guidelines define substantial risk for HIV and recommend PrEP be an option for individuals reporting: partner of HIV-infected person not on ART or on ART for <6 months, >1 partner of unknown status, transactional sex, recent STI, recurrent PEP use, inconsistent condom use, or injection drug use. So, non-pregnant cisgender women reporting any of these factors will not be eligible for the study but will be linked for PrEP at clinic of choice including at Thika Site itself.
* Willing to be randomized to non-daily PrEP and come to clinic frequently for DOT PrEP
* Willingness and ability to be abstinent for at least 7 days after each vaginal biopsy visit.

Specific for pregnant cisgender women only

* At screening, evidence of a viable pregnancy with gestational age of 13-26 weeks after the date of conception with sonographic confirmation. If adequate sonographic results are not available from medical records at screening, an ultrasound must be performed in the interim so that the result is available at study entry.
* At elevated risk for acquiring HIV according to Kenya guideline for PrEP. This is to ensure an ethical approach for provision of PrEP in pregnancy (i.e., only exposing PrEP to those who want and might benefit from it). Kenya national guidelines define substantial risk for HIV and recommend PrEP be an option for individuals reporting partner of HIV-infected person not on ART or on ART for <6 months, >1 partner of unknown status, transactional sex, recent STI, recurrent PEP use, no or inconsistent condom use
* At study entry, willing to use PrEP during pregnancy for HIV prevention

Exclusion Criteria:

* For all cisgender women
* Inability to give informed consent
* Positive screening HIV+ as determined by standard rapid serologic assays or suspected acute HIV infection in the opinion of the clinician. (example signs and symptoms of acute HIV infection include combinations of fever, headache, fatigue, arthralgia, vomiting, myalgia, diarrhea, pharyngitis, rash, night sweats, and adenopathy cervical or inguinal)
* Positive HBV surface antigen test at screening
* Calculated creatinine clearance < 60 ml/min.
* Any laboratory value or uncontrolled medical conditions that, in the opinion of the investigators, would interfere with the study conditions such as, heart disease and/or cancer.
* Prohibited concomitant medications are: investigational agents (within 30 days of enrollment), aminoglycosides, ganciclovir/valganciclovir, chronic high-dose acyclovir/valacyclovir (>800mg acyclovir or > 500mg valacyclovir for >7 days), cyclosporine, amphotericin B, foscarnet, and cidofovir, and products with same or similar active ingredients as the study medications including TAF®, ATRIPLA®, COMPLERA®, EMTRIVA®, VIREAD®; or drugs containing lamivudine or adefovir, which are close analogs of FTC and tenofovir, respectively.
* Current or past use of PrEP (pre-exposure prophylaxis)
* Not willing to have home visits

Specific for non-pregnant cisgender women cohort

* Pregnancy or plan to become pregnant in the next 6 months or unwillingness to use birth control
* Current breastfeeding
* High risk of HIV infection (for example: sexually active with an HIV infected partner; engages in condomless intercourse with HIV-infected partners or partner of unknown status during the study; females who exchange sex for money, shelter, or gifts; active injection drug use or during the last 12 months; newly diagnosed sexually transmitted infections in last 6 months.

Specific for pregnant cisgender women cohort

* Mother has a known history of any of the following, as determined by the site investigator or designee based on maternal report and available medical records:
* Sickle cell anemia (excluding sickle cell trait), chronic bleeding, blood transfusion within the past 120 days (excluding for chronic illness) or other blood dyscrasias
* Fetus has a known or suspected major congenital anomaly, from chart review of prior data, defined ultrasound.
* Complications in prior pregnancies that would be considered exclusionary

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Steady state concentrations of tenofovir-diphosphate for different dosing patterns of DOT TDF/FTC PrEP | Assessed through 8 weeks
  Measured in dried blood spots, whole blood, PBMCs
Steady state concentrations of tenofovir for different dosing patterns of DOT TDF/FTC PrEP | Assessed through 8 weeks
  Measured in plasma, whole blood, vaginal tissue
Composite outcome of adverse pregnancy outcomes among pregnant women who used DOT PrEP | Assessed at delivery (approximately through 40 weeks gestation)
  Descriptive frequency indicating presence vs. absence of any adverse pregnancy outcomes. Adverse outcomes are defined as at least one of the following: spontaneous abortion (less than 20 weeks gestation), stillbirth (greater than or equal to 20 weeks gestation), preterm delivery (less than 37 weeks), or small for gestational age (less than 10th percentile using WHO norms)

SECONDARY OUTCOMES:
Frequency of Grade 2 or higher adverse events in participants | Assessed through 8 weeks of DOT TDF/FTC PrEP
  Based on signs, symptoms, labs, and diagnoses
Frequency of infant death among infants of women in the pregnant cohort | Assessed through 12 months after delivery
  Based on safety-related data recorded on case report forms and complete expedited adverse event (EAE) reporting by site investigators
Frequency of infant Grade 2 or higher adverse events among infants of women in the pregnant cohort | Assessed through 12 months after delivery
  Assessed according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Mugwanya, MBChB, MS, PhD, Principal Investigator — University of Washington; Peter L Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kenya Medical Research Institute - Partners in Health Research and Development, Thika, Kenya

REFERENCES:
- [Derived] Mugwanya KK, Saina M, Mugo NR, MaWhinney S, Morrow M, Schaafsma TT, Donnell D, Glidden DV, Ngure K, Brown CE, Rechkina EA, Chohan BH, Wu L, Hill E, Koome E, Akelo N, Mbaire S, Morrison SA, Kibatha M, Njeru I, Muriithi M, Coppinger C, Bushman L, Baeten JM, Anderson PL; Women Benchmark Study Team. Adherence thresholds for emtricitabine-tenofovir disoproxil fumarate preexposure prophylaxis against HIV acquisition in cisgender women: A randomized directly observed dosing study. PLoS Med. 2025 Sep 9;22(9):e1004732. doi: 10.1371/journal.pmed.1004732. eCollection 2025 Sep. PMID 40924774
- [Derived] Wu L, Saina M, Brown C, Chege D, Donnell D, Glidden DV, Ngure K, Mugo NR, Akelo N, Schaafsma T, Anderson PL, Mugwanya KK. Establishing adherence-concentration-efficacy thresholds of TDF-FTC pre-exposure prophylaxis for HIV prevention in African women: a protocol for the Women TDF-FTC Benchmark Study. Front Reprod Health. 2024 May 27;6:1325257. doi: 10.3389/frph.2024.1325257. eCollection 2024. PMID 38860025